CLINICAL TRIAL: NCT04829526
Title: Firm Observational Clinical Unicenter Study on Guillain Barré Syndrome (FOCUS on GBS)
Brief Title: Firm Observational Clinical Unicenter Study on Guillain Barré Syndrome
Acronym: FOCUS on GBS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-00402; ko21Sutter
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Guillain-Barre Syndrome (GBS)
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — Retrospective extraction of demographic, clinical, laboratory, and electrophysiological data from the digital medical records

SUMMARY:
The aim of this retrospective observational single-center cohort study is to gain a deeper understanding regarding the frequency, the clinical and electrophysiologic characteristics (e.g., the diagnostic work up), complications, treatment regimes, and their associations with specific courses of disease and outcomes in adult patients with the suspected or proven diagnosis of GBS.

DETAILED DESCRIPTION:
Guillain Barré Syndrome (GBS) is a rare and life-threatening neurological emergency. The aim of this retrospective study including adult GBS patients from the last 15 years treated at the University Hospital of Basel is to assess data regarding diagnostic workup, treatment, clinical course including complications and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* suspected diagnosis of GBS, who have been treated at the University Hospital of Basel from 01.01.2005-28.02.2021

Exclusion Criteria:

* Patients with documented refusal of the general consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with the suspected and with the final proven diagnosis of GBS in the years 2005-2021
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
frequency of GBS | one time retrospective assessment at baseline
  frequency of GBS of all consecutive adult patients with the suspected initial diagnosis of GBS (admitted to the University Hospital Basel)
clinical characteristics of GBS | one time retrospective assessment at baseline
  clinical characteristics of GBS of all consecutive adult patients with the suspected initial diagnosis of GBS (admitted to the University Hospital Basel)
electrophysiologic characteristics of GBS | one time retrospective assessment at baseline
  electrophysiologic characteristics of GBS of all consecutive adult patients with the suspected initial diagnosis of GBS (admitted to the University Hospital Basel)
complications of GBS | one time retrospective assessment at baseline
  complications of GBS of all consecutive adult patients with the suspected initial diagnosis of GBS (admitted to the University Hospital Basel)
treatment regimes of GBS | one time retrospective assessment at baseline
  treatment regimes of GBS of all consecutive adult patients with the suspected initial diagnosis of GBS (admitted to the University Hospital Basel)
outcomes of GBS | one time retrospective assessment at baseline
  treatment regimes of GBS of all consecutive adult patients with the suspected initial diagnosis of GBS (admitted to the University Hospital Basel)

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, Prof. Dr. med., Principal Investigator — Clinic for Intensive Care Medicine, University Hospital Basel
Locations (1):
- Clinic for Intensive Care Medicine; University Hospital Basel, Basel, Switzerland